CLINICAL TRIAL: NCT05066555
Title: Circulating Tumor DNA Genotyping for Biological Monitoring of Patients with Advanced-stage Classical HL Receiving Upfront ABVD-based Chemotherapy. an Ancillary Study to the FIL-Rouge Phase III Trial
Brief Title: Circulating Tumor DNA Genotyping for Biological Monitoring of Patients Treated in the FIL-Rouge Clinical Trial
Acronym: FIL-RougeBIO
Status: Completed | Type: Observational
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Other Study IDs: FIL-RougeBIO
Record Dates: First submitted 2021-09-06; First posted 2021-10-04 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Hodgkin Lymphoma
Keywords: Hodgkin Lymphoma; ABVD treatment; ancillary; ctDNA; cHL; FIL-Rouge; PFS; Response Rate
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples will be collected in Cell-Free DNA BCT tubes before treatment start, at the interim PET/CT (Positron Emission Tomography/Computed Tomography), at the end of treatment assessment, and at the time of disease progression/relapse and will be analyzed for ctDNA (Circulating tumor DNA) and gDNA (genomic DNA) genotyping and for cytokines and chemokines levels.
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Advanced-stage Hodgkin Lymphoma patients (1): All patients will be accrued by investigators from the 19 best recruiting centers in the FIL-Rouge clinical trial. Patients had undergone to ABVD-based upfront treatment in FIL-Rouge trial (Comparator arm).
- Advanced-stage Hodgkin Lymphoma patients (2): All patients will be accrued by investigators from the 19 best recruiting centers in the FIL-Rouge clinical trial. Patients had undergone to ABVD-based upfront treatment in FIL-Rouge trial (Experimental arm).

SUMMARY:
Prospective, multicenter, non-interventional, biological study ancillary to FIL-Rouge clinical trial (NCT03159897) enrolling patients affected by Advanced-stage Hodgkin Lymphoma, ABVD-based upfront treatment in 19 centers in Italy part of Fondazione Italiana Linfomi.

DETAILED DESCRIPTION:
The FIL-Rouge design provides an ideal environment for validating the liquid biopsy in Classical Hodgkin lymphoma (cHL), since one arm of the study will utilize a PET/CT-adapted strategy (Positron Emission Tomography/Computed Tomography)for treatment, while the second arm will be devoid of any PET/CT-adaptation of therapy. Also, estimating prospectively differences in residual disease between the two study arms of the FIL-Rouge will provide an important biologic tool to validate the concept of dose-intensification within the ABVD therapeutic platform.

This study aims at the prospective validation of the concept of the liquid biopsy as a biomarker for disease response assessment in cHL. The patients enrolled in the FIL-Rouge clinical trial at the centers participating in this study and consenting to the biological study FIL-RougeBIO will be considered for this study. After providing written informed consent, relevant patients will be evaluated for detecting cancer gene mutations in ctDNA (Circulating Tumor DNA) for measuring residual disease. All clinical data useful for data analyses of this study will derive from the FIL-Rouge clinical trial.

Given the non-interventional design of the study, project participants will not have immediate potential benefits.The enrollment in FIL-RougeBIO will parallel the original protocol until reaching the 500 programmed patients. The results of this study could benefit future patients with the same condition.

ELIGIBILITY:
Inclusion Criteria: FIL ROUGE INCLUSION CRITERIA

* Histologically confirmed classical HL
* Previously untreated disease
* Age 18-60 years
* Ann Arbor stage IIB with extranodal involvement and/or bulk, III and IV
* At least one target PET-avid bidimensionally assessable lesion
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) <= 2
* Adequate organ and marrow function as defined below:

  * Absolute neutrophil count >1,0 x109/L, platelets >75 x109/L
  * Total bilirubin <2 mg/dl without a pattern consistent with Gilbert's syndrome
  * Aspartate Transaminase and Alanine Transaminase (AST/ALT) <3 X institutional Upper Limits of Normality (ULN)
  * Creatinine within normal institutional limits or creatinine clearance >50 mL/min/1.73 m2
* Females of childbearing must have a negative pregnancy test under medical supervision even if patients had been using effective contraception
* Life expectancy > 6 months
* Able to adhere to the study visit schedule and other protocol requirements
* Signed (or legally acceptable representatives must sign) informed consent indicating that patients understand the purpose of and procedures required for the study and are willing to participate in the study.
* Access to PET-CT (Positron Emission Tomography/Computed Tomography) scans facilities qualified by FIL

Exclusion Criteria: FIL ROUGE EXCLUSION CRITERIA

* Nodular Lymphocyte Predominant HL
* Ann Arbor stage IIB without extranodal involvement and/or mediastinal bulky
* Prior chemotherapy or radiation therapy
* Pregnant or lactating females
* Known hypertension, cardiac arrhythmia, conduction abnormalities, ischemic cardiopathy, left ventricular hypertrophy or left ventricular ejection fraction (LVEF) ≤50% at echocardiography.
* Abnormal QTc interval prolonged (>450 msec in males; >470 msec in women)
* Diffusion lung capacity for CO (DLCO)and/or Forced expiratory volume in the 1st second (FEV1) tests <50% of predicted not due to mediastinal compression or parenchymal lymphoma
* Known cerebral or meningeal disease (HL or any other etiology)
* Prior history of malignancies unless the patient has been free of the disease for five years. Exceptions include the following: basal cells carcinoma of the skin, squamous cell carcinoma of the skin, carcinoma in situ of the cervix, carcinoma in situ of the breast and prostate cancer with the TNM stage of T1a or T1b
* Uncontrolled infectious disease
* Human immunodeficiency virus (HIV) positivity or active infectious A, B or C hepatitis. HBsAg-negative patients with anti-HBc (Hepatitis B core) antibody and can be enrolled provided that Hepatitis B Virus (HBV)-DNA are negative and that antiviral treatment with nucleos(t)ide analogs is provided (Lamivudine)
* Uncompensated diabetes
* Refusal of adequate contraception
* Any medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Eligibility criteria for participation in this study require:
  * Enrollment in the FIL-Rouge clinical trial;
  * Evidence of signed informed consent for the biological FIL-RougeBIO study.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2024-11-03 (Actual)

PRIMARY OUTCOMES:
Complete Response Rate (CRR) | The endpoint will be assessed from the beginning of the study up to 76 months
  Complete Response Rate (CRR) is defined as the proportion of patients achieving a Complete Remission (CR) at the end of treatment;

SECONDARY OUTCOMES:
Diagnostic accuracy of Circulating tumor DNA (ctDNA) analysis versus interim PET/CT (Positron Emission Tomography/Computed Tomography) | The endpoint will be assessed from the beginning of the study up to 76 months
  Diagnostic accuracy of Circulating tumor DNA (ctDNA) analysis versus interim PET/CT (sensitivity, specificity, positive predictive value, negative predictive value, positive and negative likelihood ratios accuracy); The endpoint will be evaluated through specific timepoints.
Progression Free Survival (PFS) with at least three years of follow up | The endpoint will be assessed from the beginning of the study up to 76 months
  PFS is defined as the interval elapsing from randomization until lymphoma progression/relapse or death as a result of any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Pinto, MD, Principal Investigator — Dipartimento di Ematologia, Istituto Nazionale Tumori, Fondazione Pascale, IRCCS, Napoli, Italy
Locations (13):
- Italy (13):
  - Azienda Ospedaliera S.Giuseppe Moscati - S.C. Ematologia e Trapianto emopoietico, Avellino
  - IRCCS Istituto Tumori Giovanni Paolo II - U.O.C Ematologia, Bari
  - ASST Spedali Civili di Brescia - Ematologia, Brescia
  - ASST Grande Ospedale Metropolitano Niguarda - SC Ematologia, Milan
  - Istituto Nazionale Tumori - IRCCS Fondazione G. Pascale - UOC Ematologia Oncologica, Napoli
  - Presidio ospedaliero "A. TORTORA" - U.O. Onco-ematologia, Pagani
  - A.O. Ospedali Riuniti Villa Sofia-Cervello - Divisione di Ematologia, Palermo
  - IRCCS Policlinico S. Matteo di Pavia - Div. di Ematologia, Pavia
  - Ospedale S. Maria della Misericordia - Ematologia, Perugia
  - P.O. Spirito Santo di Pescara - UOS Dipartimentale - Centro di diagnosi e Terapia dei linfomi, Pescara
  - Ospedale degli Infermi di Rimini - U.O. di Ematologia, Rimini
  - Istituto Clinico Humanitas - U.O. Ematologia, Rozzano
  - A.O.U. Citta della Salute e della Scienza di Torino - S.C.Ematologia, Torino

IPD SHARING:
Plan to Share IPD: Undecided